CLINICAL TRIAL: NCT00560456
Title: Chronic Sleep Restriction and Driving in Healthy Subjects or Snorers : Interindividual Vulnerability and Recovery Factors
Brief Title: Chronic Sleep Restriction and Driving
Acronym: PRIVASOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: PREDIT Go4 (Unknown)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUBX 2006/09
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-04

CONDITIONS: Sleep Deprivation
Keywords: Age, Snoring, Driving simulator, Sleep deprivation, chronic sleep restriction, objective and subjective sleepiness
MeSH Terms: conditions — Sleep Deprivation; Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): snorers
  Interventions: Other: Chronic sleep restriction and driving simulator
- 2 (Other): healthy volonters (control)
  Interventions: Other: Chronic sleep restriction and driving simulator
- 3 (Experimental): young subjects
  Interventions: Other: Chronic sleep restriction and driving simulator
- 4 (Experimental): mature subjects
  Interventions: Other: Chronic sleep restriction and driving simulator

INTERVENTIONS:
Other: Chronic sleep restriction and driving simulator — * One night of normal sleep
  * Driving simulator
  * Night 1: night of total sleep deprivation
  * Night 2: night of sleep recovery
  * Night 1 to 5: nights of sleep restriction
  * Driving simulator after night 1 to 5
  * Night 6: night of sleep recovery
  * Driving simulator

SUMMARY:
Young subjects and patients with nocturnal respiratory disorders are frequently involved in sleep-related accidents. This study assess the impact of chronic sleep restriction (4 hr of sleep during 5 days) or total sleep deprivation in young or mature healthy subjects or snorers on simulated driving, objective and subjective sleepiness and objective and subjective cognitive performances. The effects of recovery night on these parameters are also assessed.

DETAILED DESCRIPTION:
Principal objective :

To determine whether chronic sleep restriction affects more snorers driving performances than healthy subjects' driving performances.

To determine whether chronic sleep restriction affects more young people driving performances than mature subjects' driving performances.

Secondary objective :

To determine whether chronic sleep restriction affects more snorers reaction time performance and sleepiness than non snorers subjects'.

To determine whether chronic sleep restriction affects more young people reaction time performance and sleepiness than mature subjects'.

To determine how age and snoring intensity affects the degradation of performance over the 5 days of sleep deprivation.

To determine age-related changes in the time course of sleepiness during 5 days of chronic sleep restriction.

To compare the impact of total sleep or chronic sleep restriction on driving performances according to the age and snoring intensity.

To determine recovery facilities to chronic sleep restriction according to the age and snoring intensity.

Study plan :

G2: Group of subjects:

* patients
* controls

B1: Baseline normal night:

One night of normal sleep

A2: Acute sleep deprivation:

Night 1: night of total sleep deprivation Night 2: night of sleep recovery

C6: Chronic sleep deprivation:

Night 1 to 5: nights of sleep restriction Night 6: night of sleep recovery

Experimental plan : S20 <G2> *B1 * A2 *C6

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects inclusion criteria :

* Healthy males without snoring nor subjective daytime sleepiness (Epworth <9)
* Intermediate chronotype
* Hypopnea/apnea index <5
* Periodic movement index <5
* Sleep efficiency > 85 %
* Not taking medication modifying alertness
* Mean driving distance per year 15000 km
* Regular sleep-wake schedule.

Snorers inclusion criteria :

* Snoring males without subjective daytime sleepiness (Epworth <9)
* Intermediate chronotype
* Hypopnea/apnea index <5
* Periodic movement index < 5
* Sleep efficiency > 85 %
* Not taking medication modifying alertness
* Mean driving distance per year 15000 km
* Regular sleep-wake schedule

Exclusion Criteria:

Healthy subjects exclusion criteria :

* Short or long sleeper
* Shift- or night-worker
* Sleep, mood, neurological, cardiovascular, pulmonary, endocrinological,… disorders
* Alcohol
* Consumption of illicit drugs.

Snorers exclusion criteria :

* Short or long sleeper
* Shift- or night-worker
* Mood, neurological, cardiovascular, pulmonary, endocrinological,… disorders,
* Sleep disorder except snoring
* Alcohol
* Consumption of illicit drugs.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Standard deviation from the centre of the road on driving simulator | 1 week

SECONDARY OUTCOMES:
Number of inappropriate line crossing on driving simulator Number of lapses assessed by SRTT 10 % of slowest reaction time Mean sleep latency at 6*20-minutes multi sleep latency test. Subjective sleepiness (Karolinska and VAS) Nocturnal PSG | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Philip, MD, Principal Investigator — University Hospital Bordeaux, France
Locations (2):
- France (2):
  - University Hospital Bordeaux, Groupe Hospitalier Pellegrin, Bordeaux
  - Laboratoire d'Imagerie et de Neurosciences Cognitives (LINC), Strasbourg